CLINICAL TRIAL: NCT02748837
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of ERY974, An Anti-Glypican3 (GPC3)/CD3 Bispecific Antibody, in Patients With Advanced Solid Tumors
Brief Title: A Study of ERY974 in Patient With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERY101EG
Record Dates: First submitted 2016-03-29; First posted 2016-04-22 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — bispecific antibody ERY974

ARMS (4):
- Dose escalation cohort of ERY974 (Experimental): Dose escalation (DE) will proceed with the dose level increment and the dose cohort size being guided by a safety evaluations during and at the end of each cohort. DE initially utilizes an accelerated titration design (ATD) and once the first dose limiting toxicity (DLT) is observed, DE will continue using a modified continual reassessment method (mCRM) until MTD.
  Interventions: Drug: ERY974
- Cohort expansion in gastric cancer (Experimental): Patients with GPC3 positive advanced gastric cancer or gastroesophageal junction cancer will receive ERY974 at recommended dose until disease progression.
  Interventions: Drug: ERY974
- Cohort expansion in esophageal carcinoma (Experimental): Patients with GPC3 positive advanced squamous cell esophageal carcinoma will receive ERY974 at recommended dose until disease progression.
  Interventions: Drug: ERY974
- Cohort expansion in other solid tumors (Experimental): Patients with other GPC3 positive advanced solid tumors will receive ERY974 at recommended dose until disease progression
  Interventions: Drug: ERY974

INTERVENTIONS:
Drug: ERY974

SUMMARY:
This is the open label, multicenter Phase 1 study which consists of a dose escalation to determine the maximum tolerated dose (MTD) and cohort expansion to obtain a preliminary evaluation of anti-tumor activity. ERY974 is intravenously injected to patients with Glypican 3 positive advanced solid tumors until unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with Glypican 3 positive advanced solid tumor not amenable to standard therapy or for which standard therapy is not available or not indicated
* Measurable tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Adequate bone marrow, liver, and renal function
* Adequate coagulation status

Exclusion Criteria:

* Patients with more than a single brain metastasis ( >1 cm)
* Patients with acute or chronic infection
* Major surgery within 28 days
* Pregnant or lactating women
* Patients with interstitial pneumonitis
* Patients require regular ascites/pleural effusion drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Dose escalation： MTD determination | DLT evaluation period, defined as from the first ERY974 injection until 7 days after the third injection
  Determination of dose-limiting toxicities (DLT)
Cohort expansion：Preliminary assessment of change in tumor size | From the date of informed consents obtained until disease progression: at screening , week 6,12,18 and subsequently every 3 months up to 38 months
  Anti-tumor activity will be assessed by modified Response Evaluation Criteria in Solid Tumors (mRECIST)

SECONDARY OUTCOMES:
Dose escalation： Number and severity of adverse events | Adverse events will be reported through 28 days after the last dose
Dose escalation： Plasma ERY974 concentrations | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Dose escalation：Area under curve (AUC) | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Dose escalation：terminal half-life | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Dose escalation：total clearance | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Dose escalation：volume distribution | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Dose escalation： Change in tumor size assessed by mRECIST | From the date of informed consents obtained until disease progression: at screening , week 6,12,18 and subsequently every 3 months up to 38 months
Dose escalation： Determining the recommended dose | Recommended dose will be determined after completion of DLT assessments in all dose escalation cohorts. It is estimated as 18 months after first patient enrollment.
Cohort expansion：Number and severity of adverse events | Adverse events will be reported through 28 days after the last dose
Cohort expansion ：Plasma ERY974 concentrations | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Cohort expansion ：Area under curve (AUC) | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Cohort expansion ：terminal half-life | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Cohort expansion ：total clearance | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months
Cohort expansion ：volume distribution | PK will be assessed from day 1 to day 22, day 1 to day 29, or day 1 to day 36, then every 3 weeks from day 43 until end of treatment visit, up to 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (10):
- United States (7):
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Boston, Massachusetts
  - Detroit, Michigan
  - New York, New York
  - Durham, North Carolina
  - Providence, Rhode Island
- France (2):
  - Paris
  - Villejuif
- Groningen, Netherlands